CLINICAL TRIAL: NCT07206069
Title: Telemedicine for Evaluation and Counseling of Living Kidney Donor Candidates
Brief Title: Telemedicine to Support Living Kidney Donor Candidates
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Fawaz Al Ammary, Associate Professor of Medicine, Director of Mixed Methods Research., University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UC Irvine IRB#4138; K23DK129820 (NIH)
Record Dates: First submitted 2025-09-10; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Healthy; Living Kidney Donation
Keywords: Kidney donation; Telemedicine; Education; Counseling; Decision Making, Shared; Feasibility studies; Health Services Research; Care Delivery
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care Group (Control) (Active Comparator): Participants in the standard care group will receive a recorded video education session and one in-person donor evaluation and counseling session with a nephrologist.
  Interventions: Behavioral: Standard Care (in control arm)
- Telemedicine Group (Intervention) (Experimental): Participants in the telemedicine group will receive two live telemedicine video sessions: one education session with a transplant provider and one donor evaluation and counseling session with a nephrologist.
  Interventions: Behavioral: Telemedicine Shared Decision-Making

INTERVENTIONS:
Behavioral: Standard Care (in control arm) — This Standard Care involves a recorded video education and in-person visit.
  Other Names: Control
  Arms: Standard Care Group (Control)
Behavioral: Telemedicine Shared Decision-Making — This intervention involves two live telemedicine video visits.
  Other Names: Experimental
  Arms: Telemedicine Group (Intervention)

SUMMARY:
The goal of this feasibility clinical trial is to learn if telemedicine can be used to provide education and evaluation and counseling for people who are considering living kidney donation. The study will also learn how participants improve decision-making about living kidney donation. The main questions to answer are:

* Is telemedicine a practical way to facilitate donor education and evaluation and counseling?
* Does telemedicine shared decision making help improve donor candidate decision and engagement during the donor evaluation process?

Researchers will compare standard care with a telemedicine care coordination approach.

Participants will:

- Receive either standard care or telemedicine video visits to support shared decision making.

DETAILED DESCRIPTION:
Living kidney donation provides a vital treatment option for patients with kidney failure, but many willing individuals face challenges in completing the donor evaluation and committing to donation. Donor education and counseling are essential for informed decision-making, yet these steps are often limited to in-person visits at transplant centers. This can create logistical challenges, delays, and variations in access to the living donor evaluation process. Telemedicine offers an opportunity to deliver a shared decision making approach to donor education and evaluation and counseling remotely, but its feasibility, acceptability, and impact have not been well studied.

This pilot feasibility clinical trial is designed to test whether a telemedicine care coordination can support donor decision-making and engagement during the evaluation process for living kidney donation.

Participants will be randomly assigned to one of two groups:

* Standard Care Group (Control): A recorded video education session and an in-person donor evaluation and counseling with a nephrologist.
* Telemedicine Group (Intervention): Two live telemedicine video sessions-one for education with a transplant provider and one for donor evaluation and counseling with a nephrologist.

The findings from this feasibility trial will provide important information about the practicality and acceptability of telemedicine shared decision-making for living kidney donor candidates. Generated preliminary data will inform larger trials and ultimately guide transplant practice and policy to improve decision-making, efficiency, and access to living kidney donation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Reside in the State of California
* Registered living kidney donor candidate at UC Irvine Medical Center

Exclusion Criteria:

- Individuals with a contraindication to living kidney donation (for example, heart disease, cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-10-10 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | 90 days
  Proportion of eligible participants who consent and enroll in the study, calculated as the number enrolled divided by the number of eligible participants approached.
Retention Rate | 90 days
  Proportion of enrolled participants who remain in the study through the 90-day follow-up period, calculated as the number completing final follow-up divided by the number enrolled.
Change in Decisional Conflict Measured by the Decisional Conflict Scale (DCS) | 90 days
  Decision conflict will be measured using the Decisional Conflict Scale (DCS), a 16-item validated instrument. Each item is scored from 0 (no conflict) to 100 (very high conflict), and a total score is calculated by averaging across items. Total scores therefore range from 0 to 100, with higher scores indicating worse decision conflict and greater uncertainty.

SECONDARY OUTCOMES:
Completion of Donor Education and Evaluation and Counseling | 90 days
  Completion of donor education and evaluation and counseling.
  Time to donor evaluation and counseling completion.
Intervention Acceptability | Post-telemedicine session 1 at 7 days, and telemedicine session 2 at 67 days
  Participant-reported acceptability of the telemedicine intervention will be measured using the acceptability of intervention measure. This outcome will be assessed only in the Telemedicine Intervention Arm.

CONTACTS AND LOCATIONS:
Overall Officials: Fawaz Al Ammary, MD PhD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California Irvine Medical Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data that underlie the results reported in publications will be shared. This will include baseline demographic characteristics, survey responses, and donor candidate disposition data. Data will be deposited in Dryad and accompanied by a data dictionary, study protocol, and statistical analysis plan.
Supporting Information: Study Protocol, SAP
Time Frame: Shared data will be made available at the time of publication of the primary results. Data will remain available in the Dryad repository for a minimum of 5 years.
Access Criteria: Shared data will be made available through the Dryad digital repository. Supporting materials will include a data dictionary, study protocol, and statistical analysis plan. In accordance with the NIH Data Management and Sharing Plan and UC Irvine IRB guidance, no personally identifiable information will be included. Data will be shared under a CC0 waiver, allowing other researchers to reuse the de-identified data for health, medical, or biomedical research purposes.
URL: https://datadryad.org/

REFERENCES:
- [Background] Al Ammary F, Adeyemo S, Lentine KL, Muzaale AD. Evolution of Biologically Related Living Kidney Donation in the United States from 1988 to 2022. J Am Soc Nephrol. 2024 Aug 1;35(8):1104-1106. doi: 10.1681/ASN.0000000000000424. Epub 2024 May 29. No abstract available. PMID 38809617
- [Background] Al Ammary F, Yu Y, Ferzola A, Motter JD, Massie AB, Yu S, Thomas AG, Crews DC, Segev DL, Muzaale AD, Henderson ML. The first increase in live kidney donation in the United States in 15 years. Am J Transplant. 2020 Dec;20(12):3590-3598. doi: 10.1111/ajt.16136. Epub 2020 Jul 17. PMID 32524764
- [Background] Achkar KA, Abdelnour LM, Abu Jawdeh BG, Tantisattamoa E, Al Ammary F. Evaluation and Long-Term Follow-Up of Living Kidney Donors. Adv Kidney Dis Health. 2024 Sep;31(5):400-407. doi: 10.1053/j.akdh.2024.04.003. PMID 39232610
- [Background] Al Ammary F, Bowring MG, Massie AB, Yu S, Waldram MM, Garonzik-Wang J, Thomas AG, Holscher CM, Qadi MA, Henderson ML, Wiseman AC, Gralla J, Brennan DC, Segev DL, Muzaale AD. The changing landscape of live kidney donation in the United States from 2005 to 2017. Am J Transplant. 2019 Sep;19(9):2614-2621. doi: 10.1111/ajt.15368. Epub 2019 May 3. PMID 30903733
- [Background] Al Ammary F, Motter JD, Sung HC, Lentine KL, Sharfuddin A, Kumar V, Yadav A, Doshi MD, Virmani S, Concepcion BP, Grace T, Sidoti CN, Yahya Jan M, Muzaale AD, Wolf J. Telemedicine services for living kidney donation: A US survey of multidisciplinary providers. Am J Transplant. 2022 Aug;22(8):2041-2051. doi: 10.1111/ajt.17093. Epub 2022 May 31. PMID 35575439
- [Background] Al Ammary F, Muzaale AD, Tantisattamoa E, Hanna RM, Reddy UG, Bunnapradist S, Kalantar-Zadeh K. Changing landscape of living kidney donation and the role of telemedicine. Curr Opin Nephrol Hypertens. 2023 Jan 1;32(1):81-88. doi: 10.1097/MNH.0000000000000848. Epub 2022 Oct 21. PMID 36444666
- [Background] Kim E, Sung HC, Kaplow K, Bendersky V, Sidoti C, Muzaale AD, Akhtar J, Levan M, Esayed S, Khan A, Mejia C, Al Ammary F. Donor Perceptions and Preferences of Telemedicine and In-Person Visits for Living Kidney Donor Evaluation. Kidney Int Rep. 2024 May 15;9(8):2453-2461. doi: 10.1016/j.ekir.2024.05.009. eCollection 2024 Aug. PMID 39156145